CLINICAL TRIAL: NCT01955980
Title: A Pilot Study to Investigate the Potential of Buparid/PARI SINUS Versus Budes® Nasal Spray to Avoid or Postpone Sinus Surgery in Adult Patients With Chronic Rhinosinusitis
Brief Title: Buparid/PARI SINUS Versus Budes® Nasal Spray in the Therapy of Chronic Rhinosinusitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pari Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12082.102
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Rhinosinusitis
Keywords: CRS; without polyposis
MeSH Terms: conditions — Rhinosinusitis | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buparid; Treatment A (Experimental): Buparid 1mg budesonide/2 ml nebulizer solution
  Interventions: Drug: Budesonide
- Budes; Treatment B (Active Comparator): Budes Nasal Spray 50 µg budesonide/pump
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Inhalation
  Arms: Buparid; Treatment A
Drug: Budesonide — Nasal Spray
  Arms: Budes; Treatment B

SUMMARY:
The study should create data for the selection of a clinically relevant endpoint to assess the potential of Buparid/PARI SINUS to postpone sinus surgery in patients with chronic Rhinosinusitis.

DETAILED DESCRIPTION:
The objective of this study is to analyse whether Buparid/PARI SINUS has a higher potential to avoid or postpone sinus surgery in adult patients with CRS than Standard of Care therapy with Budes® Nasal Spray. The results of this study are expected to provide estimates for a proper sample size calculation to conduct a pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed diagnosis of chronic rhinosinusitis
* Patient without alternative other than sinus surgery
* Patient's written informed consent obtained prior to any screening or study-specific procedure
* Male or female, ≥ 18 years of age
* Patient is able to undergo nasal therapy without restrictions
* Capable to correctly use the PARI SINUS device
* Capable of understanding the purpose and risk of the clinical trial
* Female patients with childbearing potential must have a negative urine pregnancy test prior to first IMP administration.
* Patient is able to participate in the study according to Investigator's opinion

Exclusion Criteria:

* Patients with cystic fibrosis
* Patients with polyposis nasi grade I-IV
* Patients with prior FESS (Functional Endoscopic Sinus Surgery)
* Pregnant or breastfeeding women
* Any active invasive bacterial, viral or fungal infection within one week prior to first investigational medicinal product (IMP) administration
* No clinically relevant abnormal parameters of vital signs, blood biochemistry or renal/hepatic function
* Unlikely to comply with visits, inhalation procedures or other measurements scheduled in the protocol
* Receipt of an investigational drug as part of a clinical trial within 4 weeks prior to first administration of IMP
* Any co-existing medical condition that in the Investigator's judgement will substantially increase the risk associated with the patient's participation in the clinical trial
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary procedures
* Drug or alcohol abuse
* End-stage malignancies
* Known hypersensitivity to Budesonide
* Patients with oral steroid therapy within the last 3 months
* Patients needing > 1 mg/day Budesonide (or steroidal equivalent) for therapy of asthma
* Patients on therapy with leukotriene-receptor antagonists, decongestants, antihistamines or antibiotics
* Patients with frequent epistaxis (> 1 episode per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Canis, MD, Principal Investigator — University Goettingen
Locations (3):
- Germany (3):
  - University Göttingen, Göttingen
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz
  - University Munich, Munich

RESULTS

PARTICIPANT FLOW:
Groups:
- Buparid; Treatment A: Buparid 1mg budesonide/2 ml nebulizer solution
  Budesonide: Inhalation Solution
Period: Overall Study
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buparid; Treatment A | Budes; Treatment B | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change of Inflammation of the Nasal Mucosa and Paranasal Sinus
Description: Inflammation of the nasal mucosa and paranasal sinus was assessed using the Lund-Mackay score based on magnetic resonance imaging. The score can take on values between 0 and 24 points, with higher values indicating more severe thickness of the mucosa or opacification. The outcome investigated is the intraindividual mean score of 2 independent raters assessing the same images.
Time Frame: Change from Baseline to week 8
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 10 | 9
score on a scale | 0 [-2 to 5.5] | -0.8 [-5.5 to 4.5]

2. Secondary Outcome: Health-specific Quality of Life
Description: Health-specific quality of life was assessed by means of the self-rated, 20-item Sino-Nasal Outcome Test (SNOT-20). The SNOT-20 total score has a (theoretical) range of 0 - 100 points, with higher scores indicating more severe impairment.
  Presented are the mean values of the SNOT-20 total score after 48 weeks minus value at day 0 (baseline).
Time Frame: change of SNOT-20 total score from baseline to week 48
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 10 | 9
score on a scale | 17.1 [5.5 to 28.7] | 22.9 [10.5 to 35.3]

3. Secondary Outcome: Nasal Obstruction
Description: Nasal obstruction was assessed using the method of rhinomanometry by measuring the positive nasal inspiratory flow (PNIF). For the assessment the subject had to inhale maximally through the nose three times and the highest value of flow rate was recorded after 4 weeks and 8 weeks of treatment.
Time Frame: 4 weeks / 8 weeks
Measure: Mean (95% Confidence Interval); unit: ml/sec
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 10 | 9
ml/sec
  Mean flow rate after 4 weeks | 542.4 [521 to 664] | 582.0 [447 to 717]
  Mean flow rate after 8 weeks | 461.5 [320 to 602] | 551.5 [408 to 694]

4. Secondary Outcome: Inflammation of the Nasal Mucosa and Paranasal Sinus
Description: Determination of the thickness of the mucosa using Magnetic Resonance Imaging
Time Frame: Changes from Baseline at Week 8
Reporting Status: Not Posted

5. Secondary Outcome: Safety Assessment
Description: Treatment-emergent adverse events
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 10 | 9
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: Each participant has been monitored for adverse events up to 48 weeks. All patients withdrawn from the study will be followed-up for AEs or SAEs for further 2 weeks or 4 weeks, respectively.
Arm/Group | Buparid; Treatment A | Budes; Treatment B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/9
Other Adverse Events (participants affected / at risk) | 5/10 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buparid; Treatment A (N=10) | Budes; Treatment B (N=9)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buparid; Treatment A (N=10) | Budes; Treatment B (N=9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT01955980/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT01955980/SAP_001.pdf